CLINICAL TRIAL: NCT00656344
Title: Cognitive Behavioral Treatment of Posttraumatic Stress Disorder Enhanced by Virtual Reality for Individuals With PTSD and Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Joann Difede, Professor of Psychology in Psychiatry, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9603000551
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Posttraumatic Stress Disorder; Substance Abuse
Keywords: PTSD; Substance Abuse; WTC attacks; Iraq War
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Cognitive behavioral treatment enhanced by virtual reality — A cognitive behavioral protocol with cognitive and behavioral techniques will be used to treat symptoms. The exposure part of the treatment will be enhanced with the use of a virtual environment.

SUMMARY:
This study is exploring the use of an intervention designed to treat PTSD in individuals with comorbid PTSD and substance abuse resulting from the attacks of September 11 or from military service in Iraq. A cognitive behavioral treatment protocol will be used to treat PTSD. The exposure component of the protocol will be enhanced with the use of virtual reality in which the client will view a virtual environment while describing their trauma.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Between the ages of 18 and 70
* Exposed to the WTC Attacks (were in towers or in the immediate area) or veterans of the Iraq War
* Diagnosed with PTSD symptoms
* Current substance abuse disorder or history of substance abuse disorder

Exclusion Criteria:

* Presence of current organic mental disorder
* Presence or history of schizophrenia, bipolar disorder or depression with psychotic features, delusional disorder
* Active suicidal ideation, intent, or plan
* Active homicidal ideation, intent, or plan
* Use of pacemaker
* Medically unstable
* History of seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
posttraumatic stress symptomatology | prior to treatment, during the treatment, immediately following treatment and 6 months after the completion of treatment

SECONDARY OUTCOMES:
substance use symptomatology | prior to treatment, during treatment, immediately following treatment, and 6 months after the completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Difede, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.patss.com